CLINICAL TRIAL: NCT00525304
Title: Optimizing Chronic Illness Self-Management for Individuals With Schizophrenia
Brief Title: A Self-Management Program for Adults With Both Schizophrenia and a Co-occurring Medical Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Richard Goldberg, PI, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00040526; R34MH078168 (NIH); DAHBR 96-BHB
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
Keywords: medical co-morbidity; diabetes; heart disease; respiratory illness
MeSH Terms: conditions — Schizophrenia; Diabetes Mellitus; Heart Diseases | interventions — Self-Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive a self-management program for chronic illness
  Interventions: Behavioral: Self-management program for chronic illness
- Usaual Care (No Intervention): Usual Care; no additional intervention

INTERVENTIONS:
Behavioral: Self-management program for chronic illness — Self-management program for chronic illness will include between 10 and 16 psychoeducational and supportive group sessions.
  Arms: 1

SUMMARY:
This study will develop and evaluate the effectiveness of a self-management program for adults living with both schizophrenia and a co-occurring medical condition.

DETAILED DESCRIPTION:
Schizophrenia is a life-long brain disorder affecting approximately 1 percent of Americans each year. Schizophrenia can be extremely disabling, causing people to hear voices, experience paranoia or hallucinations, and believe that others are controlling their thoughts. People with schizophrenia also experience increased rates of concurrent medical conditions, such as diabetes, respiratory illness, and heart disease. This can make holding a job or even caring for oneself very difficult. The purpose of this study is to develop and evaluate a self-management program for adults living with both schizophrenia and a concurrent medical condition.

Participants in this open-label study will attend 10 to 16 group sessions led by two group leaders. Group sessions will meet each week for an hour during which participants will learn new skills to help them take responsibility for the daily management of chronic medical conditions. In addition to learning how to communicate more effectively with medical providers, participants will learn about healthy eating, the importance of physical activity, addictive behaviors that can worsen health conditions, and proper use of medications. Homework will be assigned weekly for participants to review skills learned in each session. After each session, participants will complete a survey to evaluate the session's effectiveness. At the end of the study, participants will attend one additional group meeting and an individual interview to discuss the overall effectiveness of the intervention and their experiences in the group sessions. The results of this study will be used to evaluate and improve the self-management program for future use.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for schizophrenia or schizoaffective disorder
* Current documented chart diagnosis of at least one chronic medical condition
* Received clinic services for a minimum of 3 months prior to study entry
* English-speaking
* Willing to use an effective form of birth control throughout the study if sexually active

Exclusion Criteria:

* History of a serious neurological disorder or head trauma with loss of consciousness
* Diagnosed with mental retardation or dementia
* Diagnosed with end stage organ disease
* Currently receiving chemotherapy and/or radiation treatment for cancer
* Received psychiatric hospitalization less than 3 months prior to study entry date
* Blind and/or deaf
* Pregnant
* Infected with HIV with a CD4 count under 350
* Diagnosis of AIDS
* Diagnosis of anorexia
* Problematic substance use, as defined by a mental health provider
* Psychiatric instability, as defined by a mental health provider

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2007-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Health-related self-efficacy and recovery orientation | Measured at pre- and post-intervention
Medical illness self-management skills | Measured at pre- and post-intervention
Social and communication skills during interactions with health care providers | Measured at pre- and post-intervention
Physical and mental health status | Measured at pre- and post-intervention
Medical service use patterns | Measured at pre- and post-intervention

SECONDARY OUTCOMES:
Medication use | Measured throughout the study
Neurocognition | Measured at baseline
Substance abuse | Measured at pre- and post-intervention
Psychiatric symptoms | Measured at pre- and post-intervention
Amount and seriousness of related comorbidities | Measured at pre- and post-intervention
Quantitative and qualitative survey ratings | Measured throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Richard W. Goldberg, PhD, Principal Investigator — University of Maryland, College Park
Locations (1):
- Fayette Street Clinics, Baltimore, Maryland, United States